CLINICAL TRIAL: NCT07016490
Title: A Phase 1 Study to Evaluate the Safety, Pharmacokinetics and Anti-tumor Activity of SSGJ-709 in Patients With Advanced Malignant Tumors
Brief Title: A Phase 1 Study of SSGJ-709 in Patients With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Collaborators: Macquarie University, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-709-101
Record Dates: First submitted 2025-05-28; First posted 2025-06-11 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: SSGJ-709 (Experimental): In dose escalation phase, SSGJ-709 will be conducted using accelerated titration and traditional 3+3 design. Dose Escalation Level includes 5 levels, Q3W IV. During or after dose escalation, any dose level that does not exceed the MTD can be expanded.
  Interventions: Drug: SSGJ-709

INTERVENTIONS:
Drug: SSGJ-709 — A bispecific antibody targeting PD-1 and LAG-3.

SUMMARY:
This study is an open-label phase I study to evaluate the safety, pharmacokinetics, and anti-tumor activity of SSGJ-709 as a single agent in patients with advanced malignancies.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn more about a new drug called SSGJ-709 . The primary aim of this clinical trial is to test the safety of SSGJ-709 at different dose levels on patients with advanced malignant tumors. The clinical trial consists of two phases. The dose escalation phase involves the process of gradually increasing the amount of drug given to find the highest dose that is safe and effective. The dose expansion phase involves the process of giving a drug at a specific dose to a larger group of participants to further evaluate its safety and effectiveness.

Participants will:

1. Receive SSGJ-709 infusion once every 3 weeks
2. Visit the clinic once every 3 weeks for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Minimum life expectancy of 3 months;
* Eastern Cooperative Oncology Group (ECOG) Performance status (PS) score of 0-1;
* Locally advanced or metastatic malignant tumors confirmed by histopathology or cytology; preferred tumor types for enrollment include head and neck squamous cell carcinoma, non-small cell lung cancer, esophageal squamous cell carcinoma or adenocarcinoma, gastric or gastroesophageal junction adenocarcinoma, colorectal adenocarcinoma, hepatocellular carcinoma, urothelial carcinoma, and clear cell renal cell carcinoma. Subjects with other tumor types may be enrolled after discussion with the sponsor；
* Subject who have failed, or has been intolerant to standard therapy, or has been considered lack standard of care for a given tumor type, and who is not able to complete surgical resection and receive curative concurrent/sequential chemoradiotherapy；
* Having at least one measurable tumor lesion as the target lesion assessed per RECIST v1.1；
* The subject has adequate hematological and organ functions；

Exclusion Criteria:

* Presence of brainstem, meningeal metastases, spinal cord metastases or compression；
* Presence of active central nervous system (CNS) metastases；
* Subjects with pleural effusion, pericardial effusion, or ascites that are clinically symptomatic or require repeated drainage；
* Subjects with other malignant tumors within 3 years prior to screening；
* Subjects with autoimmune diseases that require systemic treatment within 2 years before screening；
* Subjects are positive for human immunodeficiency virus (HIV)；
* Prior or current presence of non-infectious pneumonia/interstitial lung disease requiring systemic therapy with glucocorticoids；
* Serious infection within 4 weeks prior to the first dose or the presence of any active infection requiring systemic anti-infective therapy.
* Having received the following treatments prior to the first dose of study treatment:

  1. Having received anti-tumor therapies such as biological agents, chemotherapy and other investigational drugs not approved for marketing within 3 weeks prior to the first dose of study treatment (Patient may be enrolled if the first dose of study treatment is more than 5 half-lives of the drug from the last anti-tumor therapy);
  2. Having received small molecule targeted antineoplastic agents (e.g., tyrosine kinase inhibitor), or palliative local therapy for non-target lesions, or non-specific immunomodulatory therapy (e.g., interleukin, interferon, thymosin, tumor necrosis factor) within 2 weeks prior to the first dose;
  3. Having received herbal medicine with an anti-tumor indication within 1 week prior to the first dose;
  4. Prior immunotherapy other than anti-PD-(L)1 therapy (Patients with prior immunotherapy against other targets may be enrolled after discussion and agreement with the sponsor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLT | 21 days
  Dose limiting toxicity
Incidence of Treatment-Emergent Adverse Events | through study completion, an average of 1 year
  TEAE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.

SECONDARY OUTCOMES:
Cmax of SSGJ-709 | through study completion, an average of 1 year
  Peak Plasma Concentration
Tmax of SSGJ-709 | through study completion, an average of 1 year
  Time to peak drug concentration
AUC0-last of SSGJ-709 | through study completion, an average of 1 year
  the area under the curve (AUC) up to the last measurable concentration
Incidence of ADA | through study completion, an average of 1 year
  Number of subjects with detectable anti-drug antibodies (ADA)
ORR | every 6 weeks after first dose, through study completion, an average of 1 year
  ORR ( objective response rate) is the proportion of subjects with complete response(CR) or partial response(PR), evaluated by the investigators per RECIST v1.1
PFS assessed by investigator per RECIST v1.1 | through study completion, an average of 1 year
  Progression-free survival (PFS) is defined as the time from the date of randomization till the first documentation of disease progression assessed by the investigator or death due to any cause (whichever occurs first).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Parsonson, Principal Investigator — Macquarie University
Locations (1):
- Southern Oncology Clinical Research Unit (SOCRU), Adelaide, Australia

IPD SHARING:
Plan to Share IPD: No